CLINICAL TRIAL: NCT01043419
Title: Sympathetic Neural Outflow During Xenon Anesthesia in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS-8-09-A-101; Eudract N°2009-012449-48 (Registry Identifier: Eudract)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sympathetic Nervous System
Keywords: Xenon Anesthesia; LENOXe™ (xénon 100 % v/v) anesthesia; Muscle Sympathetic Activity; Baroreflex reagibility
MeSH Terms: interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LENOXe™ (xénon 100 % v/v) (Experimental): Influence of LENOXe™ (xénon 100 % v/v) anesthesia on Sympathetic Nervous Activity and Security under LENOXe™ (xénon 100 % v/v) anesthesia
  Interventions: Drug: xenon

INTERVENTIONS:
Drug: xenon — Inhalational gas; dose allowed max.70 Vol.% in 30 % oxygen; the duration of the treatment will be to 30 minutes

SUMMARY:
The purpose of this study is to test the hypothesis that sympathetic neural outflow to muscles as well as a sympathetic baroreflexes are not altered during xenon anesthesia in Healthy Volunteers.

DETAILED DESCRIPTION:
Objectives for this study :

* Main Objective : Influence of Xenon anesthesia on Sympathetic Nervous Activity
* Secondary Objectives : Security under LENOXe™ (xénon 100 % v/v) anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers > 18 years and < 65 years of age
* ASA physical status I
* Legal competence
* for whom the consent form has been signed

Exclusion Criteria:

* Healthy volunteers < 18 years and > 65 years of age
* Pregnancy, lactation period or missing secure anticonvulsive therapy
* Missing legal competence
* Participation in other clinical trials
* Contraindications as mentioned on §4.3 of the SPCs of LENOXe™ (xénon 100 % v/v)
* Any medication especially of Sildenafil (Viagra®) or other potency remedy
* Existing relationship of dependency to the sponsor or the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Muscle Sympathetic Activity (MSA)and Baroreflex reagibility under Xenon Anesthesia in comparison to awake | 30 minutes

SECONDARY OUTCOMES:
Arterial blood pressure, Heart frequency, Arterial O2 and CO2 Saturation,Skin conductance,Concentration of plasma catecholamines, Angiotensin & Renin under Xenon Anesthesia in comparison to awake | In continuous during 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter KIENBAUM, PD Dr., Principal Investigator — Department of Anesthesiology, University Hospital Duesseldorf, Moorenstrasse 5, D-40225 Duesseldorf
Locations (1):
- Department of Anesthesiology; University Hospital of Duesseldorf; Moorenstrasse 5, Düsseldorf, Germany

REFERENCES:
- [Background] Neukirchen M, Hipp J, Schaefer MS, Brandenburger T, Bauer I, Winterhalter M, Kienbaum P, Werdehausen R. Cardiovascular stability and unchanged muscle sympathetic activity during xenon anaesthesia: role of norepinephrine uptake inhibition. Br J Anaesth. 2012 Dec;109(6):887-96. doi: 10.1093/bja/aes303. Epub 2012 Sep 3. PMID 22945969